CLINICAL TRIAL: NCT00546611
Title: A Phase I, Single-Centre, Open-Label, Fixed-Dose Study of the Safety and Efficacy of up- to Three-Days Application of 0.05% PEP005 Topical Gel in the Treatment of Patients With Common Wart(s) (Verruca[e] Vulgaris) on the Dorsal Hand
Brief Title: The Purpose of This Study is to Determine Whether Topical Application of PEP005 is Safe for the Treatment of Common Wart(s)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No enrolement
Sponsor: Peplin (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PEP005-019
Record Dates: First submitted 2007-10-18; First posted 2007-10-19 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Warts
Keywords: PEP005; Common Wart(s); Common warts (verruca[e] vulgaris)
MeSH Terms: conditions — Warts | interventions — 3-ingenyl angelate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Active Comparator): Three day application of 0.05% PEP005 Topical Gel to one or two common warts located on the hand.
  Interventions: Drug: PEP005

INTERVENTIONS:
Drug: PEP005

SUMMARY:
Verruca vulgaris, otherwise known as the common wart, is caused by the human papillomavirus (HPV). Common warts are generally located on the hands and feet, but can also occur elsewhere (e.g., any areas of frequent contact). Common warts have a characteristic cauliflower-like surface, are typically slightly raised above the surrounding skin and are generally diagnosed by visual inspection.The treatment of warts poses a therapeutic challenge for physicians. No single therapy has been proven effective at achieving complete remission in every patient.This study will aim to evaluate an up-to a three-day course of therapy with 0.05% PEP005 Topical Gel.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients at least 18 years of age.
* A clinically diagnosed, single common cutaneous viral wart (verruca vulgaris) on the dorsal hand.
* Written informed consent has been obtained.
* Agreement from the patient to allow photographs of the common wart(s) treatment area to be taken and used as part of the study package.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-10

PRIMARY OUTCOMES:
Safety

SECONDARY OUTCOMES:
Resolution of Common Wart(s)

CONTACTS AND LOCATIONS:
Overall Officials: Angela Smith, Study Director — Peplin Operations Pty Ltd
Locations (1):
- South East Dermatology, 1202 Creek Rd, Carina Heights, Brisbane, Queensland, Australia

REFERENCES:
- See also: Central HREC — http://bellberry.com.au